CLINICAL TRIAL: NCT06380218
Title: Evaluation of Nutritional Prevention Program for Women's Cardiovascular Health on Quality of Life (SAFE)
Acronym: SAFE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Pasteur de Lille (Other)
Responsible Party: Principal Investigator, Jean-Michel Lecerf, Principal Invesigator, Institut Pasteur de Lille
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2023-A00249-36
Record Dates: First submitted 2024-03-22; First posted 2024-04-23 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Healthy Volunteers
Keywords: Nutritional and physical activity program; Prevention; Cardiovascular health; Quality of life

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nutrional and physical activity program (Experimental): 10 collective combined workshops of nutrition and physical activity = 1 per week during 10 weeks associated to margarine consumption
  Interventions: Behavioral: Nutrional and physical activity program

INTERVENTIONS:
Behavioral: Nutrional and physical activity program — Nutritional prevention and physical activity workshops associated with a substitution of saturated and/or trans fatty acids by cis-unsaturated acids via the consumption of Primevère margarine to influence lifestyle habits, quality of life and improvement of the lipid profile of women with cardiovascular risk

SUMMARY:
The objective is to evaluate the effect of a nutritional prevention program associated with the consumption of "Primevère margarine" on the quality of life of women at risk of cardiovascular disease after 10 group coaching sessions in nutrition and physical activity.

DETAILED DESCRIPTION:
The objective is to evaluate the effect of a nutritional prevention program associated with the consumption of "Primevère margarine" on the quality of life of women aged 40 to 65 with cardiovascular risk 3 months after 10 group coaching sessions.

The nutritional prevention program includes tools and 10 collective workshops to change the life behaviours (eating habits and physical activity) by assessing :

* Food balance and diversity
* Eating behaviour and representations
* Level of knowledge in nutrition
* Level of physical activity and physical inactivity
* Physical abilities: strength, balance, flexibility, cardio respiratory endurance, recovery capacity
* Behavioural barriers and educational levers to improve women's cardiovascular health

ELIGIBILITY:
Inclusion Criteria:

* BMI > 25kg/m² and/or with a waist circumference > 88 cm
* Regularly consuming butter and/or "standard" margarine rich in saturated fatty acids

Exclusion Criteria:

* Regularly consuming "healthy" margarine enriched with omega 3 (Primevere, St Hubert ω3 ...) or with phytosterols (Pro-active)
* Consuming omega-3 rich food supplements within 3 months of inclusion
* Treated with lipid-lowering agents (statins), antidiabetic or antihypertensive drugs for less than 3 months
* Suffering of eating disorders
* Presenting a medical contraindication to the practice of physical activity
* Having previously participated in a similar prevention program
* Suffering from serious chronic diseases (cancer, serious cardiovascular history, etc.)

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-07-11 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline on quality of life of women with cardiovascular risk at 3 months after a nutritional prevention program associated with the consumption of "Primevère margarine" | At 3 months after the coaching session
  Quality of Life Questionnaire Short Form-36 validated by World Health Organization (WHO)

SECONDARY OUTCOMES:
Change from baseline on life behaviours at 3 months after a nutritional prevention program associated with the consumption of "Primevère margarine" | At 3 months after the coaching session
  Lifestyle Questionnaire : consumption of alcohol and tobacco and quality of sleeping
Change from baseline on well-being at 3 months after a nutritional prevention program associated with the consumption of "Primevère margarine" | At 3 months after the coaching session
  Visual analogue scales on changes in well-being ranging from 10 (best) to 0 (worst)
Change from baseline on stress management at 3 months after a nutritional prevention program associated with the consumption of "Primevère margarine" | At 3 months after the coaching session
  Cohen Questionnaire
Change from baseline on food behaviors at 3 months after a nutritional prevention program associated with the consumption of "Primevère margarine" | At 3 months after the coaching session
  Balance and dietary diversity questionnaire proposed by the Institut Pasteur de Lille
Change from baseline on food behaviors at 3 months after a nutritional prevention program associated with the consumption of "Primevère margarine" | At 3 months after the coaching session
  Behavioural questionnaire and food representation proposed by the Institut Pasteur de Lille
Change from baseline on food and physical activity knowledge at 3 months after a nutritional prevention program associated with the consumption of "Primevère margarine" | At 3 months after the coaching session
  Food knowledge Questionnaire (10 points) Physical Activity knowledge Questionnaire (10 points)
Change from baseline on motivation to change behaviors at 3 months after a nutritional prevention program associated with the consumption of "Primevère margarine" | At 3 months after the coaching session
  Prochaska Scale: Motivation to Change raging from "I don't want to" to "I will continue to do so" Identifying Barriers and Levers for Behaviour Change Related to Physical Activity Practice and food
Change from baseline on physical behaviors at 3 months after a nutritional prevention program associated with the consumption of "Primevère margarine" | At 3 months after the coaching session
  Ricci & Gagnon questionnaire (level of physical activity and sedentary lifestyle)
Change from baseline on recovery capacity at 3 months after a nutritional prevention program associated with the consumption of "Primevère margarine" | At 3 months after the coaching session
  The using test is :
  • Ruffier Dickson test (recovery capacity) - to calculate an index of the heart's ability to adapt to physical activity with the heart rate measurement
  This index is measured like that :
  < or = 0 : excellent 0 to 2 : very good 2 to 4 : good 4 to 6 : average 6 to 8 : weak 8 to 10 : very weak > 10 : poor adaptation
Change from baseline on static balance at 3 months after a nutritional prevention program associated with the consumption of "Primevère margarine" | At 3 months after the coaching session
  The using test is :
  • Unipodal balance (static balance) Measured in seconds
Change from baseline on flexibility at 3 months after a nutritional prevention program associated with the consumption of "Primevère margarine" | At 3 months after the coaching session
  The using test is :
  • Flexible trunk and posterior chain of lower limbs (flexibility) Measured by index ranging from 5 (the palms of the hands touch the ground) to 1 (the fingertips reach the lower shins)
Change from baseline on handgrip strengh at 3 months after a nutritional prevention program associated with the consumption of "Primevère margarine" | At 3 months after the coaching session
  The using test is :
  • Grip force (handgrip strength) Measured in kilograms
Change from baseline on lower limb strengh at 3 months after a nutritional prevention program associated with the consumption of "Primevère margarine" | At 3 months after the coaching session
  The using test is :
  • Sitting/standing on chair (lower limb strength) Measured in seconds
Change from baseline on endurance at 3 months after a nutritional prevention program associated with the consumption of "Primevère margarine" | At 3 months after the coaching session
  The using test is :
  • 6 minutes walk test (endurance) Measured in meters
Change from baseline on lipids metabolism at 3 months after a nutritional prevention program associated with the consumption of "Primevère margarine" | At 3 months after the coaching session
  Blood samples will be collected to analyse: Total cholesterol, HDL, LDL, triglycerides and erythrocyte rate ω3 and ratio ω6/ω3
Change from baseline on glucose metabolism at 3 months after a nutritional prevention program associated with the consumption of "Primevère margarine" | At 3 months after the coaching session
  Blood samples will be collected to analyse fasting blood glucose
Change from baseline on cardiovascular risk at 3 months after a nutritional prevention program | At 3 months after the coaching session
  Cardiovascular risk will be collected Cardiovascular Risk Assessment SCORE. The major variables are sexe, age, smoking status or not, blood pressure and total cholesterol
Change from baseline on BMI at 3 months after a nutritional prevention program associated with the consumption of "Primevère margarine" | At 3 months after the coaching session
  Height, (m) weight (kg) to calculate BMI
Change from baseline on waist circumference at 3 months after a nutritional prevention program associated with the consumption of "Primevère margarine" | At 3 months after the coaching session
  Waist circumference (cm)
Change from baseline on body composition at 3 months after a nutritional prevention program associated with the consumption of "Primevère margarine" | At 3 months after the coaching session
  Body composition by impedance measurement: % fat mass, % lean mass
Change from baseline on systolic and diastolic blood pressure at 3 months after a nutritional prevention program associated with the consumption of "Primevère margarine" | At 3 months after the coaching session
  Systolic and diastolic blood pressure to calculate blood pressure
Satisfaction of Primevere products | On the last coaching session - 10 weeks
  Measured by comprehension and utility of Primevere tools questionnaire and perception of Primevere Margarine

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Michel Lecerf, MD, Principal Investigator — Institut Pasteur de Lille - NutrInvest
Locations (1):
- NutrInvest - Institut Pasteur de Lille, Lille, Nord, France